CLINICAL TRIAL: NCT03262155
Title: Study of Immunity Dysfunction Induced by Extracorporeal Assistance (ECMO / ECLS)
Acronym: IMPEC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3037_IMPECstudy
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Acute Respiratory Distress Syndrome; Cardiogenic Shock
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Cardiogenic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO / ECLS: Patients hospitalized for ARDS or Cardiogenic shock with ECMO / ECLS
  Interventions: Biological: Blood test
- No ECMO / ECLS: Patients hospitalized for ARDS or Cardiogenic shock without ECMO / ECLS
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test

SUMMARY:
Study of immunosuppression biomarkers in patients with ARDS or cardiogenic shock with ECMO / ECLS, compared to patients with ARDS or cardiogenic shock without ECMO / ECLS

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient hospitalized in an intensive care unit
* Patient whose initial ARDS or Cardiogenic shock began less than 5 days before admission
* Patients hospitalized for ARDS or Cardiogenic shock with ECMO / ECLS or - Patients hospitalized for ARDS or Cardiogenic shock without ECMO / ECLS

Exclusion Criteria:

* Opposition of patient, relative or legal representative for participation in the study
* Pregnant woman
* Pre-immunodepression
* Implementation of immunosuppressive therapy such as chemotherapy, cyclophosphamide, high-dose corticosteroids (> 0.5mg / kg / day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for ARDS or Cardiogenic shock with or without ECMO / ECLS
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of immunosuppression in patients with ARDS or cardiogenic shock under ECMO / ECLS hospitalized in intensive care unit | Hour 24

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No